CLINICAL TRIAL: NCT06045143
Title: Right Ventricular Septal Versus Apical Pacing: Echocardiographic Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehdaa Adel Mosallam, Resident doctor, Assiut University
Other Study IDs: LV strain in pacemaker's
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Pacemaker DDD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apical pacing: Study LV strain with speckle Echo when lead of pacemaker on apical site
  Interventions: Device: Patients undergoing DDD pacemaker implantation
- Septal pacing: Study LV strain with speckle Echo when lead of pacemaker on septal site
  Interventions: Device: Patients undergoing DDD pacemaker implantation

INTERVENTIONS:
Device: Patients undergoing DDD pacemaker implantation — compare the effect right ventricular apical versus septal pacing on left ventricular function by deformation imaging using 2D speckle tracking echocardiography.

SUMMARY:
This study aims to compare the effect right ventricular apical versus septal pacing on left ventricular function by deformation imaging using 2D speckle tracking echocardiography.

DETAILED DESCRIPTION:
Permanent cardiac pacing is the most efficient treatment for various conduction disorders, including high-degree atrioventricular block and symptomatic sick sinus syndrome. High-burden right ventricular (RV) pacing is often tolerated for decades without overt left ventricular (LV) failure in most patients. It has been shown, however, that prolonged RV pacing reduces LV function and ultimately causes heart failure. Left ventricular ejection fraction (LVEF) may decrease in specific individuals with pacemaker implants following pacing, which is called Pacing-induced cardiomyopathy (PICM). However, pacing-induced LV dysfunction (PIVD) at milder severity levels has also been documented.RV apical pacing, the classic site for pacemaker lead implantation, results in ventricular dys-synchrony and deterioration of left ventricular (LV) function and ejection fraction, like left bundle branch block. Recently, alternative sites are arising, such as right ventricular outflow tract (RVOT) and the septum. Studies show that deformation imaging by speckle tracking echocardiography following pacemaker implantation can predict the patients at higher risk for PCIM and PIVD at long-term follow-up. Deformation imaging, or strain imaging, provides unique Information on regional and global ventricular function. Global longitudinal strain is Known to be more precise than ejection Fraction. It is now used in patients with heart failure, ischemic heart disease, and Receiving chemotherapy to detect early Changes in cardiac function before changes in ejection fraction. Speckle tracking Echocardiography for strain measurement Depends on tracking of speckles throughout the Cardiac cycle in apical 4,3, and 2 chamber Views. The software allows the elaboration of myocardial deformation in 3 spatial directions: Longitudinal, radial, and circumferential. Predicting PICM and PIVD 6 months after pacemaker implantation is possible by measuring global longitudinal strain (GLS) baseline one and six months after implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients older than 18 years with conduction disturbances necessitating pacemaker implantation and
2. who had preserved LVEF (≥50%) were presented to Assuit University Heart Center.

Exclusion Criteria:

1. Patients with impaired systolic function (LVEF <50%).
2. Ischemic heart disease.
3. Significant valvular heart disease (moderate to severe).
4. Pregnancy.
5. Poor echogenic window.
6. Patient refusal.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty-four patients with high degree AV block elicited for permanent pacemaker implantation were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Right ventricular apical versus septal pacing Echocardiographic study. | 1year
  This study aims to compare the effect right ventricular apical versus septal pacing on left ventricular function by deformation imaging using 2D speckle tracking echocardiography.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fcvm.2021.705778/